CLINICAL TRIAL: NCT05177289
Title: Evaluating the Feasibility and Efficacy of Photobiomodulation Therapy in the Prevention and Management of Chemotherapy-induced Alopecia: a Randomized Controlled Trial
Brief Title: Photobiomodulation Therapy in the Prevention and Management of Chemotherapy-Induced Alopecia
Acronym: HairLight
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021/117
Record Dates: First submitted 2021-12-09; First posted 2022-01-04 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Chemotherapy-induced Alopecia
Keywords: Photobiomodulation therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Patients allocated to the treatment group will receive scalp cooling combined with thrice weekly PBM sessions during the CTx course and until one month after the end of CTx.
  Interventions: Device: Theradome® LH80 pro; Device: Scalp cooling
- Control group (Active Comparator): Patients allocated to the control group will receive scalp cooling during their CTx course.
  Interventions: Device: Scalp cooling

INTERVENTIONS:
Device: Theradome® LH80 pro — The Theradome LH80 pro is a wearable laser helmet device, which uses red laser light to stop hair loss, thicken existing hair and stimulate the growth of new hair.
  Arms: Treatment group
Device: Scalp cooling — Scalp cooling is a standard treatment that is applied to prevent hair loss during chemotherapy.

SUMMARY:
This study aims to investigate the effectiveness of photobiomodulation therapy (PBM) in the prevention and management of chemotherapy-induced alopecia (CIA). Therefore, we hypothesize that PBMT can reduce the severity of CIA in gynecological and breast cancer patients, increasing the patient's QoL.

DETAILED DESCRIPTION:
The global cancer burden keeps rising, and the accompanied side effects remain a significant concern. This project focuses on one of such complications: chemotherapy-induced alopecia (CIA). 65% of cancer patients receiving cytotoxic drugs experience CIA, which negatively impacts their QoL, as hair loss is often associated with impaired body image and increased depression rates. Up to now, prevention of CIA is based on scalp cooling, but this treatment has a highly variable success rate. Photobiomodulation (PBM) therapy is a non-invasive form of phototherapy that utilizes visible and/or near-infrared light to trigger a cascade of intracellular reactions. PBM can be used to improve wound healing, and to reduce pain, inflammation, and edema. Research shows that PBM can stimulate hair growth by increasing the blood flow to the scalp and stimulating the catagen or telogen metabolism of the hair follicle. However, the effect of PBM on CIA has not been adequately investigated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with gynecological cancer (endometrium, cervix, ovarian or vulva) or breast cancer
* Receiving chemotherapy ((Carbo)-Taxol)
* Age ≥ 18 years
* Able to comply to the study protocol
* Able to sign written informed consent

Exclusion Criteria:

* Metastatic disease
* Pregnancy
* Active infection of the scalp
* Previous diagnosis of a hair loss condition
* Interruption of chemotherapy for more than two consecutive cycles
* Medication to stimulate hair growth (e.g., Minoxidil)
* Severe psychological disorder or dementia.
* Inability to speak and understand Dutch
* Substance abuse patients or patients with medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results as judged by the investigator
* Any condition that is unstable or could affect the safety of the patient and their compliance in the study as judged by the investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Hair thickness measurement | Baseline
  The research assistant will objectively evaluate the thickness of the hair using a micrometer screw gauge.
Hair thickness measurement | Halfway into their chemotherapy (An average of 6 weeks)
  The research assistant will objectively evaluate the thickness of the hair using a micrometer screw gauge.
Hair thickness measurement | At the final chemotherapy session (An average of 12 weeks)
  The research assistant will objectively evaluate the thickness of the hair using a micrometer screw gauge.
Hair thickness measurement | One month post chemotherapy
  The research assistant will objectively evaluate the thickness of the hair using a micrometer screw gauge.
CTCAE-score | Baseline
  The patient may grade their hair loss using the CTCAE criteria.
CTCAE-score | Halfway into their chemotherapy (An average of 6 weeks)
  The patient may grade their hair loss using the CTCAE criteria.
CTCAE-score | At the final chemotherapy session (An average of 12 weeks)
  The patient may grade their hair loss using the CTCAE criteria.
CTCAE-score | One month post chemotherapy
  The patient may grade their hair loss using the CTCAE criteria.
Hair loss evaluation | Baseline
  Both the patient and a blinded study nurse will score hair regrowth based on photographs. A score of 0 equals 'total baldness' and 10 'full scalp coverage'.
Hair loss evaluation | Halfway into their chemotherapy (An average of 6 weeks)
  Both the patient and a blinded study nurse will score hair regrowth based on photographs. A score of 0 equals 'total baldness' and 10 'full scalp coverage'.
Hair loss evaluation | At the final chemotherapy session (An average of 12 weeks)
  Both the patient and a blinded study nurse will score hair regrowth based on photographs. A score of 0 equals 'total baldness' and 10 'full scalp coverage'.
Hair loss evaluation | One month post chemotherapy
  Both the patient and a blinded study nurse will score hair regrowth based on photographs. A score of 0 equals 'total baldness' and 10 'full scalp coverage'.

SECONDARY OUTCOMES:
Quality of life score | Baseline
  The European Organization for Research and Treatment for Cancer Quality of Life Questionnaire will be used to evaluate the patients' quality of life.
Quality of life score | Halfway into their chemotherapy (An average of 6 weeks)
  The European Organization for Research and Treatment for Cancer Quality of Life Questionnaire will be used to evaluate the patients' quality of life.
Quality of life score | At the final chemotherapy session (An average of 12 weeks)
  The European Organization for Research and Treatment for Cancer Quality of Life Questionnaire will be used to evaluate the patients' quality of life.
Quality of life score | One month post chemotherapy
  The European Organization for Research and Treatment for Cancer Quality of Life Questionnaire will be used to evaluate the patients' quality of life.
Satisfaction score | Halfway into their chemotherapy (An average of 6 weeks)
  The patients will be asked to evaluate their global satisfaction with the therapeutic intervention. The patients will score their satisfaction regarding their treatment on the NRS scale 0 (totally not satisfied) to 10 (very satisfied).
Satisfaction score | At the final chemotherapy session (An average of 12 weeks)
  The patients will be asked to evaluate their global satisfaction with the therapeutic intervention. The patients will score their satisfaction regarding their treatment on the NRS scale 0 (totally not satisfied) to 10 (very satisfied).
Satisfaction score | One month post chemotherapy
  The patients will be asked to evaluate their global satisfaction with the therapeutic intervention. The patients will score their satisfaction regarding their treatment on the NRS scale 0 (totally not satisfied) to 10 (very satisfied).

OTHER OUTCOMES:
General patient-, disease-, and treatment-related information | Baseline
  General and medical information will be collected through a short patient questionnaire in order to assess intrinsic risk factors (e.g. age and smoking history). Information regarding the disease- and treatment-related risk factors will be collected through medical records (e.g., tumour type and stage).
General patient-, disease-, and treatment-related information | One month post chemotherapy
  General and medical information will be collected through a short patient questionnaire in order to assess intrinsic risk factors (e.g. age and smoking history). Information regarding the disease- and treatment-related risk factors will be collected through medical records (e.g., tumour type and stage).
Cancer relapse or recurrence | One year post chemotherapy
  The posibility of cancer relapse or recurrence will be evaluated using the patients' medical records.
Cancer relapse or recurrence | Two years post chemotherapy
  The possibility of cancer relapse or recurrence will be evaluated using the patients' medical records.
Cancer relapse or recurrence | Three years post chemotherapy
  The possibility of cancer relapse or recurrence will be evaluated using the patients' medical records.
Cancer relapse or recurrence | Four years post chemotherapy
  The possibility of cancer relapse or recurrence will be evaluated using the patients' medical records.
Cancer relapse or recurrence | Five years post chemotherapy
  The possibility of cancer relapse or recurrence will be evaluated using the patients' medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Mebis, Prof. Dr., Principal Investigator — Jessa Hospital
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

REFERENCES:
- [Derived] Claes M, Robijns J, Lambrichts L, Van Duffel S, Bulens P, Mebis J. Photobiomodulation therapy in the prevention of chemotherapy-induced alopecia in breast cancer patients: a randomized controlled trial. Lasers Med Sci. 2025 Jul 24;40(1):325. doi: 10.1007/s10103-025-04577-7. PMID 40705170